CLINICAL TRIAL: NCT06778395
Title: Therapeutic Effect of Vonoprazan Versus Dexlansoprazole in Treatment of Gastroesophageal Reflux Disease in Egyptian Patients: A Prospective Comparative Study
Brief Title: Therapeutic Effect of Vonoprazan Versus Dexlansoprazole in Treatment of Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ayman Magd Eldin Mohammad Sadek (Other Government)
Collaborators: Zagazig University (Other Government)
Responsible Party: Sponsor-Investigator, Ayman Magd Eldin Mohammad Sadek, Associate Professor of Internal Medicine, Zagazig University
Organization: Zagazig University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#745/5-Nov-2024
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Vonoprazan; Proton Pump Inhibitor; Gastroesophageal Reflux Disease
Keywords: Dexlansoprazole; gastroesophageal reflux disease; Vonoprazan
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Dexlansoprazole; 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexlansoprazole (Active Comparator): 60 mg once daily
  Interventions: Drug: Dexlansoprazole 60 mg
- Vonoprazan (Active Comparator): 20 mg twice daily
  Interventions: Drug: Vonoprazan 20 mg bid

INTERVENTIONS:
Drug: Dexlansoprazole 60 mg — once daily for 8 weeks
  Arms: Dexlansoprazole
Drug: Vonoprazan 20 mg bid — twice daily for 8 weeks
  Arms: Vonoprazan

SUMMARY:
Gastroenterologists are often hesitated about whether to use the well known PPI in treatment of GERD or the usage of new H/K ATPase inhibitors so its highly needed to test the benefit of each class in Egyptian population to help doctors in decision making

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a common gastrointestinal disorder that occurs when gastric contents reflux into the esophagus and oral cavity, resulting in troublesome symptoms and/or complications. These include heartburn, a burning sensation in the chest, acid regurgitation, or an ongoing cough. Serious complications include dysphagia and Barrett's esophagus, potentially leading to esophageal adenocarcinoma.

GERD is a common condition, often due to abnormalities in the lower esophageal sphincter, with a pooled global prevalence of 13.3% or more of the population reporting at least weekly symptoms with rates increasing; however, with appreciable geographical variation. As a result, GERD is typically the most frequent gastrointestinal disorder across countries, with consultation rates in ambulatory care ranging from 5.4% to 56% of all consultations. Although GERD cannot be classified as a single disease, it is often used as an umbrella term.

Endoscopy is used to identify GERD, as well as clinical signs including heartburn and acid regurgitation. The two types of GERD are either erosive or non-erosive reflux disease.

The main therapeutic option for GERD is proton pump inhibitors [PPIs], which are superior to other medications in terms of symptom alleviation and mucosal healing. PPIs are known as first-line treatments in individuals with GERD.

Dexlansoprazole, which is the seventh proton pump inhibitor (PPI) to enter the market, is currently one of six PPIs available. It has been used clinically in various formulations as a racemic mixture. The chemical structure of lansoprazole contains an asymmetric sulfinyl group with a chiral center, resulting in two enantiomers, R (+) and S (-). Dexlansoprazole is the R-enantiomer. While the R and S isomers exhibit comparable pharmacological characteristics, research conducted in laboratory settings and living organisms has revealed that the dominant factor behind the inhibitory effects of racemic lansoprazole on the secretion of gastric acid is mainly dexlansoprazole.

Vonoprazan is known as a new family in the suppression of gastric acid which is a potassium-competitive acid blocker [P-CABs]. In comparison to PPIs, P-CABs reversibly inhibit H+ and K+ ATPase, resulting in a great and long-term suppression of acid secretion. As reported in some studies, the rate of healing of reflux esophagitis was superior to that of a PPI [lansoprazole], with a greater effect seen in cases with greater severity.

P-CABs act faster than PPIs and reach their peak in acid inhibition impact post-treatment, whereas PPIs take three to five days. However, few researchers have looked at whether Vonoprazan's faster affects the clinical impact on GERD symptoms of acid regurgitation as weak as heartburn.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of GERD through upper endoscopy

Exclusion Criteria:

* Patients with a history of previous GERD surgery
* Patients on any proton pump inhibitors (PPIs) or H2 blockers within 4 weeks prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Symptom relief assessed by the GERD-Q score | 8 weeks

SECONDARY OUTCOMES:
Frequency scale of the symptoms of gastroesophageal reflux disease questionnaire (FSSG) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Sadek, MD, Study Chair — Zagazig University
Locations (1):
- Zagazig University Hospital, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheng Y, Liu J, Tan X, Dai Y, Xie C, Li X, Lu Q, Kou F, Jiang H, Li J. Direct Comparison of the Efficacy and Safety of Vonoprazan Versus Proton-Pump Inhibitors for Gastroesophageal Reflux Disease: A Systematic Review and Meta-Analysis. Dig Dis Sci. 2021 Jan;66(1):19-28. doi: 10.1007/s10620-020-06141-5. Epub 2020 Feb 24. PMID 32095968
- [Result] Zhang M, Xiao Y, Chen M. The role of vonoprazan in patients with erosive esophagitis. Therap Adv Gastroenterol. 2022 Sep 13;15:17562848221122623. doi: 10.1177/17562848221122623. eCollection 2022. PMID 36117573
- [Result] Manabe N, Joh T, Higuchi K, Iwakiri K, Kamiya T, Haruma K, Nakada K. Clinical significance of gastroesophageal reflux disease with minimal change: a multicenter prospective observational study. Sci Rep. 2022 Sep 3;12(1):15036. doi: 10.1038/s41598-022-19408-w. PMID 36057730
- [Result] Eusebi LH, Telese A, Cirota GG, Haidry R, Zagari RM, Bazzoli F, Ford AC. Systematic review with meta-analysis: risk factors for Barrett's oesophagus in individuals with gastro-oesophageal reflux symptoms. Aliment Pharmacol Ther. 2021 May;53(9):968-976. doi: 10.1111/apt.16321. Epub 2021 Mar 11. PMID 33705573
- [Result] Turshudzhyan A, Samuel S, Tawfik A, Tadros M. Rebuilding trust in proton pump inhibitor therapy. World J Gastroenterol. 2022 Jun 28;28(24):2667-2679. doi: 10.3748/wjg.v28.i24.2667. PMID 35979162
- [Result] Richter JE, Rubenstein JH. Presentation and Epidemiology of Gastroesophageal Reflux Disease. Gastroenterology. 2018 Jan;154(2):267-276. doi: 10.1053/j.gastro.2017.07.045. Epub 2017 Aug 3. PMID 28780072
- [Result] Jung HK, Tae CH, Song KH, Kang SJ, Park JK, Gong EJ, Shin JE, Lim HC, Lee SK, Jung DH, Choi YJ, Seo SI, Kim JS, Lee JM, Kim BJ, Kang SH, Park CH, Choi SC, Kwon JG, Park KS, Park MI, Lee TH, Kim SY, Cho YS, Lee HH, Jung KW, Kim DH, Moon HS, Miwa H, Chen CL, Gonlachanvit S, Ghoshal UC, Wu JCY, Siah KTH, Hou X, Oshima T, Choi MY, Lee KJ; Korean Society of Neurogastroenterology and Motility. 2020 Seoul Consensus on the Diagnosis and Management of Gastroesophageal Reflux Disease. J Neurogastroenterol Motil. 2021 Oct 30;27(4):453-481. doi: 10.5056/jnm21077. PMID 34642267
- [Result] Al-Marhabi A, Hashem A, Zuberi BF, Onyekwere C, Lodhi I, Mounir M, Alkhowaiter S, Al Awadhi S, Naidoo VG, Hamada Y. The views of African and Middle Eastern Gastroenterologists on the management of mild-to-moderate, non-erosive gastro-esophageal reflux disease (GERD). Expert Rev Gastroenterol Hepatol. 2022 Mar;16(3):217-233. doi: 10.1080/17474124.2022.2043744. Epub 2022 Feb 25. PMID 35184616